CLINICAL TRIAL: NCT04557631
Title: Evaluation of the Threshold for the Interpretation of the Results of a Method for the Blood Determination of Phosphatidyléthanol
Acronym: PETHOXICO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_02; 2019-A02683-54 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For an analytical validation of the method for the determination of blood hosphatidylethathanol, it is necessary to:

* to compare the results of chronic and excessive ethanol patients with the cut-off proposed in the literature.
* Also assess the stability of phosphatidylethanol in total blood collected, and in blotted dried blood stains (DBS), depending on temperature (ambient temperature and +4°C)

ELIGIBILITY:
Inclusion Criteria:

* Person with alcohol consumption ≥ 40g/day (women) and ≥ 60g/day (men) according to WHO criteria
* Person hospitalized for a hospital withdrawal in the addiction service of Lille's hospital, without other distinctions.

Exclusion Criteria:

* Patient opposing the use of their personal data in the study
* Patient subject to protective measures (guardianship or curatorship)
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study will be proposed to all major ethanol-consuming patients with an alcohol use disorder, seen in consultation, in anticipation of hospital withdrawal in addiction service.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of patients with a Peth concentration greater than 200 µg/L | at the end of study (at 6 months)

SECONDARY OUTCOMES:
the concentration of Peth in blood in ambiant temperature | between T0 and 96h and the end of study (at 6 months)
  descrease expressed as a percentage of the initial concentration, in the primary blood tube (citrate tube) and stored at room temperature,
the concentration of Peth in blood at 4°C | between T0 and 96h and the end of study (at 6 months)
  ecrease expressed as a percentage of the initial concentration, in the primary blood tube (citrate tube) and at 4°C.
the concentration of Peth in blood in DBS | between T0 and 4 weeks and the end of study (at 6 months)
  decrease expressed as a percentage of the initial concentration, in the Dried Blood Spot (DBS)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, MD,PhD, Principal Investigator — University Hospital, Lille